CLINICAL TRIAL: NCT00817544
Title: Excretion Balance and Metabolism After a Single Oral Dose of 14C-Labelled ORM-12741; an Open, Non-Randomised, Single Centre Study in Healthy Male Subjects
Brief Title: Excretion Balance and Metabolism After a Single Oral Dose of 14C-Labelled ORM-12741
Acronym: ALMAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Orion Corporation, Orion Pharma (Leena Lehtonen, Clinical study director), Orion Corporation, Orion Pharma
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3098004
Record Dates: First submitted 2008-12-23; First posted 2009-01-06 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Healthy Male Volunteers
Keywords: 3098004; Healthy volunteers
MeSH Terms: interventions — ORM-12741

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ORM-12741 (Experimental): ORM-12741
  Interventions: Drug: ORM-12741

INTERVENTIONS:
Drug: ORM-12741 — 3 mg of ORM-12741 as a single dose. Contains 0.73 mg (2.5 MBq) 14C labelled ORM-12741
  Other Names: healthy volunteer

SUMMARY:
The study is conducted to examine absorption of C14-ORM-12741 from intestine to bloodstream, distribution to bloodstream, metabolism in the liver and excretion of the parent drug and metabolites to faeces, urine and expired air

DETAILED DESCRIPTION:
Six healthy males will receive 3 mg of ORM-12741 as a single oral solution(0.1mg/mL). The oral dose contains 0.73 mg of 14C-ORM-12741 (2.5 MBq), 1 mg of 13C-ORM-12741 and 1.27 mg of ORM-12741.

Subjects will be confined to the study site from Day -1 (the afternoon prior to the day of dosing) up to at least 168 hours following drug administration (Day 8). Subjects will be discharged on Day 8 if radioactivity in urine and faeces meet pre-defined criteria (urinary excretion <0.5% and faecal excretion <0.5% of the dose per 24 hours based on 14C radioactivity quick counts, which will be measured from Day 7 onwards). If on Day 8 these pre defined criteria are not met, subjects will remain hospitalised for a maximum of seven more days (Day 15) until the criteria are met (daily check on quick counts). If on Day 15 these pre defined criteria are not met, subjects will be discharged and requested to collect a 24-hour sample of urine and/or faeces at home once per week and to deliver this to the clinical research unit in Zuidlaren. These weekly collections will be continued until the criteria are met. The total duration of the study will be approximately 5 - 6 weeks for each subject.

ELIGIBILITY:
Inclusion Criteria:

* Gender male
* Age 18-60 years, inclusive
* Weight 55-100 kg, inclusive
* Body mass index (BMI) 18.0 - 30.0 kg/m2 (inclusive)
* Ability and willingness to abstain from alcohol, tobacco products, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, "power drinks"), and grape fruit (juice) from 48 hours prior to entry in the clinical research centre until discharge
* Medical history without major pathology
* All values for haematology and for clinical chemistry tests of blood and urine within normal range or showing no clinically relevant deviations as judged by the Medical Investigator
* Willingness to use adequate contraception from the time of dosing until three months after the end-of-study visit
* Willingness to sign the written Informed Consent Form (ICF)

Exclusion Criteria:

* Evidence of clinically relevant pathology
* Mental handicap
* History of relevant drug and/or food allergies
* At screening visit, abnormal 12-lead ECG of clinical relevance
* Regular/routine treatment with non-topical medication within 30 days prior to drug administration
* Irregular defecation pattern (less than once per two days)
* Exposure to radiation for diagnostic reasons (except dental X-days and plain X-rays of thorax and body skeleton (excluding spinal column)) during work or during participation in a medical trial in the previous year

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The excretion balance of total 14C-radioactivity after a single oral dose of 14C-ORM-12741 | Total 14C-radioactivity in faeces and urine until pre-defined criteria are met. The total duration of the study will be approximately 5 - 6 weeks for each subject.

SECONDARY OUTCOMES:
To gain further information on the safety of ORM-12741 | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jaap van Lier, Principal Investigator — PRA International, The Netherlands
Locations (1):
- PRA International, AE Zuitlaren, Netherlands